CLINICAL TRIAL: NCT00061776
Title: A Randomized, Double-Blind, Controlled Dose Finding Study of NGX-4010 for the Treatment of Postherpetic Neuralgia
Brief Title: NGX-4010 for the Treatment of Postherpetic Neuralgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NeurogesX (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: C108
Record Dates: First submitted 2003-06-03; First posted 2003-06-04 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-03

CONDITIONS: Herpes Zoster; Neuralgia; Pain; Peripheral Nervous System Diseases; Shingles
Keywords: Dermal assessment; Pain measurement; Diary; Shingles; Neuropathy; Analgesics/*therapeutic use; Capsaicin/*administration & dosage/adverse effects; Herpes Zoster/*complications/drug therapy; Neuralgia/*drug therapy/etiology; Pain; Peripheral Nervous System Diseases/*complications
MeSH Terms: conditions — Herpes Zoster; Neuralgia; Pain; Peripheral Nervous System Diseases

INTERVENTIONS:
Drug: Capsaicin Dermal Patch

SUMMARY:
The purpose of the study is determine if an investigational drug, NGX-4010 (high-concentration capsaicin dermal patches) is effective in treating pain associated with post-herpetic neuralgia (PHN).

DETAILED DESCRIPTION:
Participants will be randomly assigned to receive initial treatment according to one of three doses (application durations), and will receive either NGX-4010 patch (high-concentration capsaicin) or matching control (low-concentration capsaicin).

Participants who complete the study evaluations for 12 weeks will have the option of receiving up to 3 additional open-label re-treatments over 1 year.

ELIGIBILITY:
Key Eligibility Criteria:

* Must be diagnosed with PHN and be at least 6 months after crusting of the skin vesicles, with moderate to severe pain.
* Must not have significant pain due to causes other than PHN (for example, arthritis).
* Painful areas should not be located on the face, above the hairline of the scalp, and/or in proximity to mucous membranes.
* Must have intact and unbroken skin at the treatment area.
* Must be prepared to remain on the same pain medications at the same doses as before the study for the entire duration of the study (1-year).
* Must not have any implanted medical device (spinal cord stimulator, intrathecal pump or peripheral nerve stimulator) for the treatment of pain.
* Must not use topical pain medications for PHN.
* Must be able to comply with study requirements such as completing a daily pain diary, attending study visits and refraining from extensive travel during study participation.
* No significant medical problems of the heart, kidneys, liver or lungs, or cancer.
* No history or current problem with substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - NeurogesX Investigational Site, Huntsville, Alabama
  - NeurogesX Investigational Site, Phoenix, Arizona
  - NeurogesX Investigational Site, Scottsdale, Arizona
  - NeurogesX Investigational Site, Tucson, Arizona
  - NeurogesX Investigational Site, Little Rock, Arkansas
  - NeurogesX Investigational Site, La Jolla, California
  - NeurogesX Investigational Site, San Francisco, California
  - NeurogesX Investigational Site, Denver, Colorado
  - NeurogesX Investigational Site, Melbourne, Florida
  - NeurogesX Investigational Site, Naples, Florida
  - NeurogesX Investigational Site, Ocala, Florida
  - NeurogesX Investigational Site, Palm Beach Garden, Florida
  - NeurogesX Investigational Site, Plantation, Florida
  - NeurogesX Investigational Site, Sarasota, Florida
  - NeurogesX Investigational Site, St. Petersburg, Florida
  - NeurogesX Investigational Site, Boston, Massachusetts
  - NeurogesX Investigational Site, Kansas City, Missouri
  - NeurogesX Investigational Site, Las Vegas, Nevada
  - NeurogesX Investigational Site, Morristown, New Jersey
  - NeurogesX Investigational Site, Albany, New York
  - NeurogesX Investigational Site, Rochester, New York
  - NeurogesX Investigational Site, Eugene, Oregon
  - NeurogesX Investigational Site, Memphis, Tennessee
  - NeurogesX Investigational Site, Austin, Texas
  - NeurogesX Investigational Site, Dallas, Texas
  - NeurogesX Investigational Site, San Antonio, Texas
  - NeurogesX Investigational Site, Salt Lake City, Utah
  - NeurogesX Investigational Site, Tacoma, Washington